CLINICAL TRIAL: NCT02854722
Title: Phase 2 Study of Deferasirox-calcium-vitamin D3 to Treat Postmenopausal Osteoporosis (PMOP)
Brief Title: The Deferasirox-calcium-vitamin D3 Therapy for Postmenopausal Osteoporosis (PMOP)
Acronym: PMOP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, You-Jia Xu, Director of Science and Education Department, Second Affiliated Hospital of Soochow University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BL2014044
Record Dates: First submitted 2016-07-19; First posted 2016-08-03 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Postmenopausal Osteoporosis
Keywords: deferasirox; iron accumulation
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Deferasirox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deferasirox and calcium-vitamin D3 (Experimental): Deferasirox is an orodispersible tablet and should be taken daily 30 minutes before breakfast, with a dose of 10 mg/Kg/day ± 5 mg/Kg/day during 12 month.
  Calcium 500 mg and Vitamin D3 800 IU should also be taken daily as a basic therapy.
  Interventions: Drug: Deferasirox and calcium-vitamin D3; Drug: Calcium-vitamin D3
- Calcium-vitamin D3 (Placebo Comparator): Calcium 500 mg and Vitamin D3 800 IU are taken daily as a basic therapy.
  Interventions: Drug: Calcium-vitamin D3

INTERVENTIONS:
Drug: Deferasirox and calcium-vitamin D3 — deferasirox and calcium-vitamin D3 Deferasirox is an orodispersible tablet and should be taken daily 30 minutes before breakfast, with a dose of 10 mg/Kg/day ± 5 mg/Kg/day during 12 month.
  Calcium 500 mg and vitamin D3 800 IU should also be taken daily as a basic therapy.
  Arms: Deferasirox and calcium-vitamin D3
Drug: Calcium-vitamin D3 — Calcium 500 mg and vitamin D3 800 IU are taken daily as a basic therapy.

SUMMARY:
In 2006, Weinberg proposed a hypothesis that iron accumulation was a risk factor for osteoporosis. Osteoporosis is a common complication in various diseases, such as hemochromatosis, African hemosiderosis, thalassemia, and sickle cell disease, which all share iron accumulation as a common denominator. Moreover, a 3-year retrospective longitudinal study has shown that iron accumulation was also associated with osteoporosis in healthy adults and especially that it can increase the risk of fractures in postmenopausal women. Based on these observations, iron chelation therapy may have a promising future in the treatment of iron accumulation-related osteoporosis by removing iron from the body.

The purpose of this study is to determine whether the addition of the iron chelator, deferasirox, to standard therapy for postmenopausal osteoporosis, is safe and effective.

DETAILED DESCRIPTION:
Postmenopausal osteoporosis (PMOP) is a systemic bone metabolism disease, characterized by progressive bone loss following menopause and a subsequent increase in fracture risk. Estrogen deficiency as a result of menopause is known to increase bone resorption and accelerate bone loss. Furthermore, postmenopausal women may exhibit iron accumulation, in addition to estrogen deficiency. Elevated iron levels are a risk factor for PMOP in postmenopausal women, and reducing the iron overload by iron chelators has been demonstrated to benefit bone cell metabolism in vitro and improve the bone in vivo by normalizing osteoclastic bone resorption and formation.

Although the safety and efficacy of deferasirox have been evaluated in iron-overloaded patients extensively, there are no data in iron-accumulated postmenopausal women, let alone in iron-accumulated postmenopausal women with osteoporosis. Therefore, at the currently planned dose, confirming safety and efficacy is essential in the current study to lay the groundwork for a future phase III clinical trial.

This is a prospective, phase II, randomized, open label, placebo-controlled study of calcium-vitamin D3 plus deferasirox vs. calcium-vitamin D3 for postmenopausal osteoporosis. Ten postmenopausal women diagnosed with osteoporosis by DXA, who were accompanied by iron accumulation (serum 500ng/ml≤ferritin≤1000ng/ml), will be randomized to receive calcium-vitamin D3 plus deferasirox or calcium-vitamin D3 (n = 5 per arm).

The primary objective is to determine the safety and tolerability of adjunctive deferasirox therapy in postmenopausal women being treated with calcium-vitamin D3 for osteoporosis, and to obtain exploratory data on the efficacy of the iron chelation treatment. The reduction in iron levels with deferasirox may provide a viable therapeutic option for mitigating the iron accumulation associated with PMOP.

ELIGIBILITY:
Inclusion Criteria:

1. Lumbar spine or hip BMD T-score ≤-2.5 SD.
2. Elevated serum ferritin (females: serum 500ng/ml≤ferritin≤1000ng/ml).

Exclusion Criteria:

1. Anemia < 10 g/dl
2. Serum liver enzymes or bilirubin above the upper limit of normal at screening.
3. Patients with creatinine clearance <60 ml/min will be excluded.
4. Known allergy or contraindication to the administration of Deferasirox.
5. History of blood transfusion during the 6 months prior to study entry.
6. Oral iron supplementation within the last 4 weeks of study entry.
7. Treatment with phlebotomy within 2 weeks of screening visit.
8. Patient is already taking deferasirox therapy for any reason at the time of screening.
9. Patients currently or previously treated with deferiprone or Deferasirox.
10. Patients with active inflammatory diseases that may interfere with the accurate measurement of serum ferritin.
11. Patients with a diagnosis of a clinically relevant cataract or a previous history of clinically relevant ocular toxicity related to iron chelation.

Ages: 60 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-01-15 (Actual); Primary Completion 2019-06-15 (Estimated); Study Completion 2020-06-15 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events | 12 months
  An adverse event was any untoward medical occurrence in participants, and did not necessarily need to have a causal relationship with the drug in the trial. The relationship of each adverse event to study drug or the severity of each adverse event was judged by the investigator, as described below. A serious adverse event is an adverse event occurring at any dose that resulted in any of the following outcomes or actions:
  fatal or life-threatening; requires inpatient hospitalization; persistent or significant disability/incapacity;
Number of participants with abnormal blood pressure, heart rate, body temperature, and/or physical examination that are related to the treatment | 12 months
Bone mineral density | Baseline, Month 6, Month 12
  Bone mineral density was measured by dual energy X-ray absorptiometry (DXA) scan. Percent changes in DXA Bone Mineral Density from baseline to month 6 and month 12 of the trial in all patients. Percent change from Baseline was calculated as (BMD at Month 6 or Month 12 - BMD at Baseline)/BMD at Baseline * 100%.

SECONDARY OUTCOMES:
Change from baseline in serum C-terminal telopeptide of type I collagen (β-CTX) | Baseline, Month 3, Month 6, Month 9 and Month 12
Change from baseline in serum N-aminoterminal prepeptide of type I procollagen (P1NP) | Baseline, Month 3, Month 6, Month 9 and Month 12
Change from baseline in serum ferritin | Baseline, Month 3, Month 6, Month 9 and Month 12
Change from baseline in blood chemistry | Baseline, Week 2, Week 4 and Month 3, Month 6, Month 9, Month 12 of the trial
Change from baseline in hematology | Baseline, Week 2, Week 4 and Month 3, Month 6, Month 9, Month 12 of the trial

CONTACTS AND LOCATIONS:
Overall Officials: You-Jia Xu, Ph.D,M.D., Principal Investigator — Second Afflilated Hospital of Soochow University
Locations (1):
- Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kim BJ, Ahn SH, Bae SJ, Kim EH, Lee SH, Kim HK, Choe JW, Koh JM, Kim GS. Iron overload accelerates bone loss in healthy postmenopausal women and middle-aged men: a 3-year retrospective longitudinal study. J Bone Miner Res. 2012 Nov;27(11):2279-90. doi: 10.1002/jbmr.1692. PMID 22729843
- [Background] Mitchell F. Bone: high body iron stores lead to bone loss. Nat Rev Endocrinol. 2012 Sep;8(9):506. doi: 10.1038/nrendo.2012.127. Epub 2012 Jul 17. No abstract available. PMID 22801718
- [Background] Li GF, Pan YZ, Sirois P, Li K, Xu YJ. Iron homeostasis in osteoporosis and its clinical implications. Osteoporos Int. 2012 Oct;23(10):2403-8. doi: 10.1007/s00198-012-1982-1. Epub 2012 Apr 14. PMID 22525981
- [Background] Huang X, Xu Y, Partridge NC. Dancing with sex hormones, could iron contribute to the gender difference in osteoporosis? Bone. 2013 Aug;55(2):458-60. doi: 10.1016/j.bone.2013.03.008. Epub 2013 Mar 22. No abstract available. PMID 23523718
- [Background] Chen B, Yan YL, Liu C, Bo L, Li GF, Wang H, Xu YJ. Therapeutic effect of deferoxamine on iron overload-induced inhibition of osteogenesis in a zebrafish model. Calcif Tissue Int. 2014 Mar;94(3):353-60. doi: 10.1007/s00223-013-9817-4. Epub 2014 Jan 12. PMID 24414856
- [Background] Chen B, Li GF, Shen Y, Huang XI, Xu YJ. Reducing iron accumulation: A potential approach for the prevention and treatment of postmenopausal osteoporosis. Exp Ther Med. 2015 Jul;10(1):7-11. doi: 10.3892/etm.2015.2484. Epub 2015 May 8. PMID 26170904
- [Background] Shen GS, Yang Q, Jian JL, Zhao GY, Liu LL, Wang X, Zhang W, Huang X, Xu YJ. Hepcidin1 knockout mice display defects in bone microarchitecture and changes of bone formation markers. Calcif Tissue Int. 2014 Jun;94(6):632-9. doi: 10.1007/s00223-014-9845-8. Epub 2014 Mar 21. PMID 24652331
- [Background] Xu Y, Li G, Du B, Zhang P, Xiao L, Sirois P, Li K. Hepcidin increases intracellular Ca2+ of osteoblast hFOB1.19 through L-type Ca2+ channels. Regul Pept. 2011 Dec 10;172(1-3):58-61. doi: 10.1016/j.regpep.2011.08.009. Epub 2011 Sep 10. PMID 21911012
- [Background] Jia P, Xu YJ, Zhang ZL, Li K, Li B, Zhang W, Yang H. Ferric ion could facilitate osteoclast differentiation and bone resorption through the production of reactive oxygen species. J Orthop Res. 2012 Nov;30(11):1843-52. doi: 10.1002/jor.22133. Epub 2012 May 8. PMID 22570238